CLINICAL TRIAL: NCT00265564
Title: Effectiveness of Screening and Treatment for PTSD in SUD Patients
Brief Title: SUPER Study (Substance Use and PTSD Treatment Effectiveness Research Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 04-175
Record Dates: First submitted 2005-12-13; First posted 2005-12-14 (Estimated); Results first posted 2020-09-07 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-08

CONDITIONS: Substance Use Disorders; Posttraumatic Stress Disorder
Keywords: outcomes assessment; substance use disorders; stress disorders, post-traumatic; screening
MeSH Terms: conditions — Substance-Related Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Seeking Safety (Active Comparator): Seeking Safety is a manualized, empirically supported, cognitive behavioral therapy that treats substance use disorders and comorbid PTSD. Participants assigned to the Seeking Safety arm attend two one hour sessions of group therapy for 12 weeks.
  Interventions: Behavioral: Modified Seeking Safety integrated into std outpatient SUD care
- Usual Care (Active Comparator): Usual Care Condition. Patients randomized to usual care will receive standard outpatient SUD treatment.
  Interventions: Behavioral: Standard outpatient SUD care

INTERVENTIONS:
Behavioral: Modified Seeking Safety integrated into std outpatient SUD care — The Seeking Safety treatment involves two (one hour) sessions of manualized group therapy for 12 weeks.
  Other Names: Seeking Safety
  Arms: Seeking Safety
Behavioral: Standard outpatient SUD care — Patients assigned to standard care meet twice weekly in "Recovery 1" groups, which focuses on building abstinence.
  Arms: Usual Care

SUMMARY:
This study proposes a prospective program of research that will identify feasible and inexpensive methods to detect and treat comorbid PTSD among VA SUD patients, thereby improving substance abuse treatment outcomes.

DETAILED DESCRIPTION:
Background: This study proposes a prospective program of research that will identify feasible and inexpensive methods to detect and treat comorbid PTSD among VA SUD patients, thereby improving substance abuse treatment outcomes.

Objective(s): Our objectives are to test the effectiveness of substituting 2 hours/week of Seeking Safety-based groups for standard substance use focused groups for male patients attending outpatient substance use disorder treatment who meet clinical criteria for PTSD. Primary outcomes measures will assess substance use disorder severity and secondary outcome measures will assess mental health and substance use related problems plus treatment satisfaction. We hypothesize that enhanced SUD treatment that incorporates "Seeking Safety" will improve SUD treatment outcomes for PTSD-SUD patients as compared to outcomes for PTSD-SUD patients receiving treatment as usual. Additionally, we examine two hypothesized models via which "Seeking Safety" may effect substance use outcomes. We examine whether 1) reductions in PTSD symptomatology and 2) improvements in coping strategies used in response to PTSD symptoms (reductions in using to cope and other avoidance coping strategies) partially mediate the effect of treatment on substance use outcomes.

Methods: This is a randomized clinical trial of 210 male veterans with PTSD and substance use disorders attending outpatient substance use disorder treatment at the VA Oakland mental health center. Patients will be randomized to 3 months of outpatient substance abuse treatment including either 2 hours/week of "Seeking Safety" or standard addiction focused group therapy. Data will be collected in patient interviews at treatment entry and at 3, 6 and 12 months after treatment initiation and by medical record review. Substance use, PTSD symptomatology, mental health, social functioning, legal problems, use of coping techniques, and treatment satisfaction outcomes will be assessed at treatment entry and 3, 6 and 12 months later using well-validated survey instruments. Primary and secondary treatment outcomes of patients in "Seeking Safety" versus treatment as usual will be compared by repeated measures ANCOVA. We will test the mediational hypotheses according to the 4-step method described by Baron and Kenny (1986).

Status: Project began in January, 2006; Recruitment, treatment and assessment is complete and primary trial finds are published. Secondary analysis is ongoing.

ELIGIBILITY:
Inclusion Criteria:

1. veteran status and VA healthcare eligibility,
2. a diagnosis of any alcohol or drug use disorder,
3. having completed an intake for outpatient SUD treatment at the VA Oakland outpatient mental health clinic, and
4. meeting criteria for a PTSD diagnosis based on a preliminary screen with the PC-PTSD and subsequent full clinical evaluation using the CAPS

Exclusion Criteria:

1. current participation in any day or inpatient mental health treatment,
2. any contraindications communicated by that patient's primary clinician,
3. acute psychosis, mania, dementia, or suicidal intent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2006-07 (Actual); Primary Completion 2011-04 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jodie A. Trafton, PhD, Principal Investigator — VA Palo Alto Health Care System
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

REFERENCES:
- [Result] Weaver CM, Trafton JA, Walser RD, Kimerling RE. Pilot test of seeking safety treatment with male veterans. Psychiatr Serv. 2007 Jul;58(7):1012-3. doi: 10.1176/ps.2007.58.7.1012. No abstract available. PMID 17602023
- [Result] Boden MT, Kimerling R, Jacobs-Lentz J, Bowman D, Weaver C, Carney D, Walser R, Trafton JA. Seeking Safety treatment for male veterans with a substance use disorder and post-traumatic stress disorder symptomatology. Addiction. 2012 Mar;107(3):578-86. doi: 10.1111/j.1360-0443.2011.03658.x. PMID 21923756
- [Result] Oliva EM, Harris AH, Trafton JA, Gordon AJ. Receipt of opioid agonist treatment in the Veterans Health Administration: facility and patient factors. Drug Alcohol Depend. 2012 May 1;122(3):241-6. doi: 10.1016/j.drugalcdep.2011.10.004. Epub 2011 Nov 23. PMID 22115887
- [Result] Midboe AM, Cucciare MA, Trafton JA, Ketroser N, Chardos JF. Implementing motivational interviewing in primary care: the role of provider characteristics. Transl Behav Med. 2011 Dec;1(4):588-94. doi: 10.1007/s13142-011-0080-9. PMID 24073081
- [Result] Harris AH, Oliva E, Bowe T, Humphreys KN, Kivlahan DR, Trafton JA. Pharmacotherapy of alcohol use disorders by the Veterans Health Administration: patterns of receipt and persistence. Psychiatr Serv. 2012 Jul;63(7):679-85. doi: 10.1176/appi.ps.201000553. PMID 22549276
- [Result] Tyler Boden M, Kimerling R, Kulkarni M, Bonn-Miller MO, Weaver C, Trafton J. Coping among military veterans with PTSD in substance use disorder treatment. J Subst Abuse Treat. 2014 Aug;47(2):160-7. doi: 10.1016/j.jsat.2014.03.006. Epub 2014 Apr 13. PMID 24854218
- [Result] Zimmerman L, Lounsbury DW, Rosen CS, Kimerling R, Trafton JA, Lindley SE. Participatory System Dynamics Modeling: Increasing Stakeholder Engagement and Precision to Improve Implementation Planning in Systems. Adm Policy Ment Health. 2016 Nov;43(6):834-849. doi: 10.1007/s10488-016-0754-1. PMID 27480546
- [Result] Kearney LK, Smith C, Kivlahan DR, Gresen RC, Moran E, Schohn M, Trafton J, Zeiss AM. Mental health productivity monitoring in the Veterans Health Administration: Challenges and lessons learned. Psychol Serv. 2018 Nov;15(4):486-495. doi: 10.1037/ser0000173. Epub 2017 Jul 17. PMID 28714721

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Seeking Safety | Usual Care
Started | 59 | 58
Completed | 49 | 49
Not Completed | 10 | 9
Not completed — Lost to Follow-up | 5 | 7
Not completed — met exclusion criteria | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Seeking Safety | Usual Care | Total
Number analyzed (Participants) | 49 | 49 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.30 (9.38) | 53.01 (9.96) | 54.13 (9.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 49 | 49 | 98
Region of Enrollment [Number; unit: participants]
  United States | 49 | 49 | 98

OUTCOME MEASURES:

1. Primary Outcome: Severity of Alcohol Use (ASI Alcohol Composite Scores)
Description: Alcohol and drug use composite scores were separately analyzed. The ASI alcohol composite score measures the severity of substance use and amount of use in the past 30 days and consequences of use. Scored as values between 0 and 1 with higher values indicating more severe substance use (i.e. lower values indicate a better outcome).
Time Frame: Administered at baseline and 3 months, 6 months and 12 months post baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Seeking Safety | Usual Care
Number analyzed (Participants) | 49 | 49
units on a scale
  Baseline | .259 (.264) | .225 (.237)
  3 months | .169 (.191) | .152 (.129)
  6 months | .138 (.173) | .141 (.146)
  12 months | .149 (.168) | .134 (.137)
Statistical Analysis 1: Comparison: Seeking Safety vs Usual Care; We investigated treatment condition differences in change of drug and alcohol use over four time-points using generalized linear mixed modeling analyses. A trajectory for each participant was modeled yielding estimates of baseline scores (intercept), slope, and error. Four between-person parameters were estimated: average baseline score for all participants, average slope over time in TAU condition, effect of being in SS on average intercept, effect of being in SS on average slope; Test type: Superiority or Other; p > .05, Mixed Models Analysis

2. Primary Outcome: ASI Drug Composite Score
Description: Addiction Severity Index (ASI) drug composite scores measure past 30 days substance use (McLellan et al., 1992). The ASI assesses lifetime and current use of all major classes of drugs of abuse, history of substance-related problems, and history of SUD treatment. Scored as values between 0 and 1 with higher values indicating more severe substance use (i.e. lower values indicate a better outcome).
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Seeking Safety | Usual Care
Number analyzed (Participants) | 49 | 49
units on a scale
  Baseline | .089 (.080) | .106 (.084)
  3 months | .057 (.062) | .095 (.091)
  6 months | .051 (.060) | .088 (.091)
  12 months | .046 (.053) | .066 (.062)
Statistical Analysis 1: Comparison: Seeking Safety vs Usual Care; Test type: Superiority; p < .05, Mixed Models Analysis

3. Secondary Outcome: PTSD Symptoms (IES Total Score)
Description: Composite measures of PTSD symptoms. Items are rated on a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). Total score ranging from 0 (not at all) to 88 (extremely)
Time Frame: Administered at 3 months, 6 months and 12 months post enrollment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Seeking Safety | Usual Care
Number analyzed (Participants) | 49 | 49
units on a scale
  Baseline | 46.76 (19.49) | 47.66 (16.26)
  3 months | 40.80 (20.86) | 42.40 (21.30)
  6 months | 38.90 (16.72) | 36.47 (16.94)
  12 months | 35.26 (20.44) | 34.07 (17.72)
Statistical Analysis 1: Comparison: Seeking Safety vs Usual Care; Generalized linear mixed modeling analysis; Test type: Superiority or Other; p > .05, Mixed Models Analysis

ADVERSE EVENTS:
Arm/Group | Seeking Safety | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/49
Other Adverse Events (participants affected / at risk) | 0/49 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes